CLINICAL TRIAL: NCT03102268
Title: Exosomes-derived ncRNAs As Biomarkers In Cholangiocarcinoma Patients
Brief Title: ncRNAs in Exosomes of Cholangiocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: EXO-CN-1607
Record Dates: First submitted 2017-03-08; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Cholangiocarcinoma; Benign Biliary Stricture
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cholangiocarcinoma patients: cholangiocarcinoma patients without any anti-cancer therapy
- benign biliary stricture patients: benign biliary stricture patients without any therapy targeting the stricture

SUMMARY:
Exosomes are part of extracellular vesicles(EVs), and can be secreted into the environment by many types of cells. It has been demonstrated that the content and function of exosomes depends on the originating cell and the conditions under which they are produced.Exosomes contain proteins,RNAs and lipid,which may transfer biological information and activities from donor cells to receptor cells. Non-coding RNAs are involved in many biological activities including tumor growth and metastasis.

In this prospective translational study, preclinical and clinical phases have been designed. On the first step, the main goal is to characterize the ncRNAs of cholangiocarcinoma derived exosomes. This exosome biomarker may provide a useful diagnostic tool. As a second step, the study will evaluate the prognostic and predictive value of cholangiocarcinoma exosomes levels in plasma in a prospectively recruited cohort of cholangiocarcinoma patients before and after surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* 1.Provide signed informed consent. The subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign informed consent, approved by the Independent Ethic Committee (IEC)/Institutional Review Board (IRB) prior to the initiation of any study-specific procedures.

  2.Men or women aged >= 18 years. 3.Histology- or imaging-confirmed bile duct stricture. 4.Metastatic disease or locally advanced disease not amenable to curative surgery.

  5.Radiographically assessable, non-measurable disease or measurable disease as per RECIST criteria.

  6.Life expectancy of at least 8 weeks from the time of enrollment. 7.No other malignancy within the past 5 years. 8.No prior chemotherapy for advanced disease.

Exclusion Criteria:

- 1.Pregnant or lactating females. 2.Significant neurological or psychiatric disorders (psychotic disorders, dementia or seizures) that would prohibit the understanding and giving of informed consent.

3.Active Hepatitis B or C or history of an HIV infection. 4.Active uncontrolled infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be adults with cholangiocarcinoma and benign biliary stricture, candidates to receive a first-line systemic therapy, who meet all of the inclusion criteria and none of the exclusion criteria within 28 days prior to the first day of study treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of the ncRNAs | Up to 3 years from start of study
  Characterization of the ncRNAs in tumor derived exosomes from cholangiocarcinoma patients before anti-cancer therapies and benign biliary stricture patients

SECONDARY OUTCOMES:
Overall survival | Up to 3 years from start of the study
  Correlation of exosomes-derived ncRNAs(at baseline and monthly during therapy until death) and time-to-event end-points
Progression-free survival | Up to 3 years from start of the study
  Correlation of exosomes-derived ncRNAs(at baseline and monthly during therapy until tumor progression) and time-to-event end-points

CONTACTS AND LOCATIONS:
Overall Officials: Lin Miao, MD, Principal Investigator — Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ge X, Tang L, Wang Y, Wang N, Zhou J, Deng X, Zhong Y, Li Q, Wang F, Jiang G, Miao L. The diagnostic value of exosomal miRNAs in human bile of malignant biliary obstructions. Dig Liver Dis. 2021 Jun;53(6):760-765. doi: 10.1016/j.dld.2020.11.010. Epub 2020 Nov 27. PMID 33257140